CLINICAL TRIAL: NCT00737178
Title: A Randomized Trial of Immediate Versus Delayed Insertion of the Copper T380A Following Medication Abortion
Brief Title: Immediate Versus Delayed Insertion of the Copper Intrauterine Device (IUD) After Medication Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Anne Davis, Associate Professor of OBGYN, Family Planning, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAD0438
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Contraception
Keywords: IUD; Intrauterine device; Intrauterine contraception; Medication abortion; Medical abortion
MeSH Terms: interventions — Intrauterine Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate IUD insertion (Active Comparator): Insertion of CuT380A at the routine medication abortion follow-up visit one week after initiation of a medication abortion
  Interventions: Device: CuT380A
- Delayed IUD insertion (Active Comparator): Insertion of CuT380A four to six weeks after initiation of a medication abortion
  Interventions: Device: CuT380A

INTERVENTIONS:
Device: CuT380A — Comparison of different timing of IUD insertion
  Other Names: IUD, Copper T

SUMMARY:
After medication abortion, women may quickly become pregnant again and therefore need an effective birth control method right away. Intrauterine devices (IUDs) are very effective for preventing pregnancy. IUDs are usually placed more than a month after abortion. This study will randomly assign women having a medication abortion to two groups, either having the IUD inserted one week after medication abortion or having the IUD inserted more than four weeks later. Women will be followed for six months to compare how many return for IUD placement in the two groups, how many are using the IUD after six months, experience with pain, bleeding, and cramping, how easy or difficult it is to insert the IUD, how many IUDs are expelled or removed, and how many women are using any birth control six months after the abortion.

DETAILED DESCRIPTION:
Women presenting for medication abortion are highly motivated to initiate contraception and are also at high risk for repeat pregnancy. Intrauterine devices (IUDs) are among the most effective reversible methods. IUD insertion is routinely planned for at least four weeks after medication abortion. This leaves women vulnerable to pregnancy while waiting for IUD placement, and many will not return for this visit. While immediate IUD insertion after surgical abortion is known to be safe and effective, it has not been studied after medication abortion.

This study will recruit women undergoing medication abortion at Special Gynecology Services who desire an IUD for contraception. Women will be randomized to two groups: immediate insertion of the copper IUD at the routine one week follow up visit, or delayed insertion of the copper IUD at least four weeks after the medication abortion.

The primary objective of this study is to compare six month IUD prevalence between the immediate and delayed IUD insertion groups. Secondary outcomes include comparison of IUD insertion rates, continuation rates, expulsion and removal rates, and use of any contraception at six months. Pain experienced during insertion and provider ease of insertion will be recorded. A diary collected for four weeks following medication abortion will reveal the impact of early IUD placement on bleeding and cramping. Lastly, we will correlate endometrial stripe thickness and IUD position to outcomes of interest: continuation, expulsion, and removal rates.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing medication abortion
* 18 or older
* Desires IUD as birth control method for a minimum of six months
* Speaks Spanish or English
* Has a working phone number or pager
* Is willing to attend visits and will be in the area for next six months
* Has signed informed consent

Exclusion Criteria:

* Chlamydia, gonorrhea, or pelvic inflammatory disease within the past three months
* Known bleeding diathesis including anti-coagulation
* Uterine abnormality including sub-mucous myomas that significantly distort the uterine cavity
* Current cervical, uterine, or ovarian malignancy
* high-grade squamous intraepithelial lesion on most recent pap
* IUD insertion contraindicated by the World Health Organization's Medical Eligibility Criteria for Contraceptive Use (category 3 or 4)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Davis, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Special Gynecology Services, New York, New York, United States

REFERENCES:
- [Result] Shimoni N, Davis A, Ramos ME, Rosario L, Westhoff C. Timing of copper intrauterine device insertion after medical abortion: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):623-628. doi: 10.1097/AOG.0b013e31822ade67. PMID 21860292
- [Result] Shimoni N, Davis A, Westhoff C. Can ultrasound predict IUD expulsion after medical abortion? Contraception. 2014 May;89(5):434-9. doi: 10.1016/j.contraception.2014.01.006. Epub 2014 Jan 18. PMID 24560483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women presenting to Columbia University's Special Gynecology Services for medication abortion will receive comprehensive contraceptive counseling. Those interested in the Intrauterine Device (IUD) for contraception will be offered study participation. Those who accept enrollment in the study and sign consent will be randomized into 1 of 2 groups.
Pre-assignment Details: For both groups, the routine 1 week follow-up visit will confirm a successful medication abortion by passage of gestational sac on sonogram. Endometrial stripe thickness will be also be noted. For both groups a transvaginal sonogram will be performed immediately after IUD insertion to confirm IUD position.
Groups:
- Immediate IUD Insertion: IUD insertion at the routine medication abortion follow-up visit one week after initiation of a medication abortion
- Delayed IUD Insertion: IUD insertion four to six weeks after initiation of a medication abortion
Period: Overall Study
Arm/Group | Immediate IUD Insertion | Delayed IUD Insertion
Started | 71 | 85
Completed | 66 | 76
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate IUD Insertion | Delayed IUD Insertion | Total
Number analyzed (Participants) | 71 | 85 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 85 | 156
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 85 | 156
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 71 | 85 | 156

OUTCOME MEASURES:

1. Secondary Outcome: Insertion Rates
Description: Insertion rates are the proportion of women in each allocation group (immediate, delayed) who ultimately had the IUD inserted within the 6 month study period.
Time Frame: By six months after medication abortion
Measure: Number; unit: participants
Arm/Group | Immediate IUD Insertion | Delayed IUD Insertion
Number analyzed (Participants) | 71 | 85
participants | 69 | 65
Statistical Analysis 1: Comparison: Immediate IUD Insertion vs Delayed IUD Insertion; Test type: Superiority or Other; p < .01, Chi-squared

2. Secondary Outcome: Expulsion and Removal Rates
Description: Expulsion rates were defined as the number of IUDs expelled from the uterus among participants who had the IUD inserted during the study.
  Removal rates were defined as the number of IUDs that were electively removed by participant request among participants who had the IUD inserted during the study.
Time Frame: Within six months of medication abortion
Population: Per protocol: insertion and removal rates were calculated only for participants undergoing IUD insertion
Measure: Number; unit: participants
Arm/Group | Immediate IUD Insertion | Delayed IUD Insertion
Number analyzed (Participants) | 69 | 65
participants
  Expulsions | 8 | 7
  Removals | 10 | 5

3. Primary Outcome: Use of the IUD for Contraception at Six Months
Description: Six months after enrollment, we determined whether or not women were using the IUD through in-person exit interviews and phone interviews. This was an intention to treat analysis, comparing the proportion of women using the IUD based on their group assignment (immediate or delayed).
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Immediate IUD Insertion | Delayed IUD Insertion
Number analyzed (Participants) | 71 | 85
participants | 49 | 51
Statistical Analysis 1: Comparison: Immediate IUD Insertion vs Delayed IUD Insertion; Test type: Superiority or Other; p = 0.24, Chi-squared

ADVERSE EVENTS:
Arm/Group | Immediate IUD Insertion | Delayed IUD Insertion
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/85
Other Adverse Events (participants affected / at risk) | 0/71 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes